CLINICAL TRIAL: NCT07226609
Title: A Decentralized Randomized Dietary Trial in Newly Diagnosed Multiple Myeloma - NUTRIVENTION5
Brief Title: A Dietary Study for People With Multiple Myeloma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Blood Cancer United (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-237
Record Dates: First submitted 2025-11-04; First posted 2025-11-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Dietary Trial; Dietary Risk Factors; High fiber plant-based diet; 25-237
MeSH Terms: conditions — Multiple Myeloma | interventions — Nutrition Policy; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: This is a nontherapeutic study testing a high fiber plant based dietary intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (UC) (Active Comparator): Usual care (UC) While receiving standard induction chemotherapy as part of routine care, participants will have phone calls with a member of the study team every 4 weeks. At the end of standard induction chemotherapy, participants will have a phone call or video call with a dietitian.
  Interventions: Other: dietary guidelines, research dietitian visit; Behavioral: Questionnaires
- Intervention arm (Experimental): While receiving standard induction chemotherapy as part of routine care,participants will have a phone call or video call with a dietitian every 2 weeks for 12 weeks and will receive high-fiber plant-based meals for 12 weeks.
  Interventions: Other: nutrition counseling and coaching; Behavioral: Questionnaires; Other: Frozen pre-prepared meals

INTERVENTIONS:
Other: nutrition counseling and coaching — In addition to individual counseling, patients will be able to join optional group sessions every 2 weeks as well as text message check-ins for survey completion reminders. Patients will receive 12 frozen, fixed pre-made lunch and dinner shipped to their home weekly from Modify Health for 12 weeks.
  Arms: Intervention arm
Other: dietary guidelines, research dietitian visit — Participants will have phone calls with a member of the study team every 4 weeks as well as text message check-ins for survey completion reminders. At the end of standard induction chemotherapy, participants will have a phone call or video call with a dietitian
  Arms: Usual care (UC)
Behavioral: Questionnaires — Block FFQ survey, EORTC QLQ C30 survey, EORTC MY20 survey, Pre intervention survey, Post intervention survey
Other: Frozen pre-prepared meals — Patients will receive 12 frozen, fixed pre-made lunch and dinner shipped to their home weekly from Modify Health for 12 weeks.
  Arms: Intervention arm

SUMMARY:
The purpose of the study is to find out whether a dietary intervention can affect treatment response and/or quality of life for people with newly diagnosed multiple myeloma receiving standard induction chemotherapy with daratumumab (or isatuximab), lenalidomide, bortezomib, and dexamethasone (DRVd). The researchers will measure quality of life by having participants complete questionnaires. The study will investigate the effects of diet on quality of life, treatment response, and other disease, microbiome, and immune markers.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed multiple myeloma
* Patients must have pathologically confirmed multiple myeloma on bone marrow biopsy with cytogenetics via Florescence in Situ Hybridization (FISH) or SNP array or genomic sequencing report and evaluation of blood myeloma markers (quantitative immunoglobulins, free light chains, serum protein electrophoresis and immunofixation).
* Age ≥ 18 years
* Bone marrow involvement
* Planned for four 28-day cycles of daratumumab (or isatuximab), lenalidomide, bortezomib, dexamethasone (or any other steroid) (DRVd) induction chemotherapy (with once weekly bortezomib day 1, 8, 15 and lenalidomide 21/28 days).
* All 4 planned drugs initiated by C2D1.
* Must enroll before C1D21 of induction chemotherapy as study intervention starts at C2D1.
* Treatment at a site where treating oncologist has capability and plan to send for bone marrow MRD negativity by next generation sequencing at end of 4 cycles (EOI). To be confirmed with local oncologist at enrollment.
* Treatment at MSK or at a site that uses EPIC for electronic medical records and willing to share records with MSK through EPIC's Care Everywhere or through MSK's shared care network.
* Enrollment on another trial that allows for 4 cycles of 28-day DRVd is acceptable.
* Prior dexamethasone treatment is eligible.
* Patients who have received up to one cycle of cyclophosphamide and/or bortezomib with dexamethasone for disease control are eligible.
* Able to complete study procedures and visits.
* Patients on GLP-1 drugs are eligible if it has been started at least 3 months prior to C2D1 DRVd or if it has been started more recently for diabetes mellitus control but not weight loss. If it is medically indicated and started for diabetes mellitus control while on trial they will not be removed/excluded from trial.
* Participant or caregiver must be able to complete surveys.
* Baseline 24-hour dietary recall must consume <30 grams dietary fiber per day to be eligible.
* Patients that already follow a minimally processed (whole food) plant-based diet in the last 3 months are not eligible (ovo-lacto-vegetarian or processed junk food vegan diets are eligible).

Exclusion Criteria:

* Leptomeningeal/CNS involvement
* Prior cycles of combination cytotoxic infusion chemotherapy such as VDPACE or DCEP are not eligible.
* Patients with BMI ≤19 kg/m2 are excluded.
* If in the opinion of the investigator there maybe any concerns regarding the ability of the patient to complete the study safely or any contraindications.
* Severe allergy to any legume (such as anaphylactic shock) or allergies to multiple legumes or if cross-contamination is a risk are not eligible.
* Severe allergies such as anaphylactic shock to peanuts and/or tree nuts, such as cashews are not eligible.
* Enrollment onto concurrent therapeutic study that requires patient receives treatment other than 4 cycles of DRVd induction as described above.
* Concurrent weight loss or dietary programs will be ineligible if require a specific diet or weight loss supplements.
* Plan for prolonged travel during the study that would preclude adherence to prescribed diet. Willingness to comply during travel is not an exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease negative complete response (MRD-CR) rate | 1 year
  rates by IMWG criteria

SECONDARY OUTCOMES:
compare the rates of improvement in QOL | 1 year
  global health status per EORTC QLQ C30 survey administration

CONTACTS AND LOCATIONS:
Overall Officials: Urvi A Shah, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/